CLINICAL TRIAL: NCT01294904
Title: Studies of Infertility in Patients With Chronic Kidney Disease
Brief Title: Mechanisms of Infertility and Hormonal Changes in Patients With Chronic Kidney Disease
Status: Withdrawn | Type: Observational
Why Stopped: Not active
Sponsor: Lund University (Other)
Responsible Party: Sponsor
Other Study IDs: CKD and infertility
Record Dates: First submitted 2011-01-21; First posted 2011-02-14 (Estimated); Last update posted 2018-12-21 (Actual); Status verified 2018-12

CONDITIONS: Infertility
Keywords: Hormone; Sperm; Chronic kidney disease
MeSH Terms: conditions — Infertility; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Samples are stored at SUS, Malmö, Sweden
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- renal transplant patients: Patients undergoing transplantation
- dialysis patients: hemodialysis patients and peritoneal dialysis patients. Before and after a dialysis session
- patients with renal insufficiency: outpatient patients with chronic kidney disease stage 2, 3 and 4
- Chronic kidney disease: outpatient cohort. Those with mild renal insufficiency

SUMMARY:
Patients with chronic kidney disease (both men and women), especially those with terminal renal failure, manifest infertility. There has been demonstrated several hormonal changes in patients on dialysis. Increased levels of luteinizing hormone (LH) has been seen in men (12). In women the opposite has been reported. The number of spermatocytes is reduced and a disturbance in maturation has been observed.

This project is aimed to study the influence of uremic milieu on fertility in men and women. The hypopituitary/hypothalamus gland axis and hormonal levels will be studied.

DETAILED DESCRIPTION:
Renal elimination of hormones and peptides. By using a human transplantation model the investigators will study changes in hormonal levels before and after a successful transplantation up to 12 months. Hormones: testosterone, SHBG (sex hormone binding globulin), LH (luteinizing hormone), FSH (follicle stimulating hormone), estradiol and inhibin B.

Analysis of sperm quality, concentration, motility, morphology and as well DNA-fragmentation index (DFI) in men with chronic kidney disease. In women the investigators will study the maturation of follicles via vaginal ultrasound. Controls are persons from a study at Dept of Reproductive Medicine.

ELIGIBILITY:
Inclusion Criteria:

* GFR-levels

Exclusion Criteria:

* > 50 years old

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: outpatient cohorts
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-01; Primary Completion 2017-05 (Actual); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
concentration of sex hormone levels in plasma | up to three years

SECONDARY OUTCOMES:
sperm motility | up to three years

CONTACTS AND LOCATIONS:
Overall Officials: Anders Christensson, MD, Principal Investigator — Lund University
Locations (2):
- Sweden (2):
  - Dag Eckersten, Malmo
  - SUS, Malmö, Sweden, Malmo